CLINICAL TRIAL: NCT06156345
Title: Additional Effect of Forward Head Posture Correction on Temporomandibular Dysfunction: A Randomized Controlled Trial.
Brief Title: Additional Effect of Forward Head Posture Correction on Temporomandibular Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shima Abdollah Mohammad Zadeh (Other)
Responsible Party: Sponsor-Investigator, Shima Abdollah Mohammad Zadeh, Principal Investigator, University of Sharjah
Organization: University of Sharjah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Added FHP correction on TMD
Record Dates: First submitted 2023-11-24; First posted 2023-12-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Temporomandibular Disorder; Forward Head Posture
Keywords: Temporomandibular dysfunction; Pain; Traction; conservative treatment
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Permuted block randomization to ensure an equal number of allocations in each of the three groups (Conservative only and conservative with Denneroll cervical traction orthodontic). Each random block was stored in opaque sealed envelopes consecutively numbered with a third researcher. Once each participant officially joins the study the researcher will open the subsequent envelop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative (Active Comparator): consists of teaching the patient the relaxed jaw position and stretching exercises for masseter and pterygoid muscles with hold of 20-30 seconds and 3-5 repetitions. In addition to placebo traction.
  Interventions: Other: Conservative
- Conservative with Denneroll (Experimental): Participants will be supine lining with the orthotic will be placed under participants' neck.
  Treatment session time begin with 3 minutes then increase of 2-3 minutes until they reach 15 to 20 minutes in each session with the conservative management for TMD.
  Interventions: Device: Conservative with Denneroll

INTERVENTIONS:
Device: Conservative with Denneroll — Denneroll cervical traction orthodontic traction for 3 to 15 minutes once daily with conservative management of stretching and relaxation.
  Arms: Conservative with Denneroll
Other: Conservative — conservative management of stretching and relaxation with placebo traction.
  Arms: Conservative

SUMMARY:
The goal of this clinical trial is to test the additional correction effect of nerd neck on damaged jaw in people who suffers from jaw problems and nerd neck at the same time. The main question it aims to answer:

• whether the additional correction of nerd neck impact the jaw features of pain and function.

Participants will:

* participants will be given the consent to sign first.
* participants will be assessed to check jaw pain and function.
* participants will be divided randomly into 2 groups.
* Each group will be given the treatment sessions for 6 weeks.
* participants will come back after 6 weeks for another last assessment. Researchers will compare regular treatment for Jaw with new device, regular only and dental treatment groups to see if there is improvement in jaw characteristics.

DETAILED DESCRIPTION:
The relationship between the two conditions of forward head posture (FHP) and temporomandibular joint dysfunction (TMD) have been previously stated with comparing the craniocervical angle (CVA) of TMD patients to the healthy individuals, still a clear relationship couldn't be drawn due to different study limitations such as the lack of subdivision in the TMD patients based on their diagnostic subcategories in addition to, patients' posture might have been altered while the photo was captured. Ever since, multiple researchers deliberately investigated the two conditions association and inferred the following: 1. FHP can be a risk factor resulting in TMD where any alteration in the head position produces more tension on the masticatory muscles by changing the mandible position 2. TMD origins from muscular component is more significant than articular component yet the correlation between head posture and TMD is still not clear enough, however, if FHP and myogenic TMD were linked preventive measures can be taken. recently, multiple studies established a relation between the occurrence of FHP in TMD patients which supported the suspected relation between them but without a clear association. Till present, no study has investigated the additional effect of FHP DCTO correction impact on myogenic TMD, and this is where the purpose of this study arises from.

ELIGIBILITY:
Inclusion Criteria:

* The participant experiencing one or more of TMD signs or symptoms and has been diagnosed with TMD beside having forward head posture with craniocervical (CVA) angle < 50.
* The study will be limited to the patients in the dental clinic of the university of Sharjah.
* Participants experiencing mild to moderate myogenic TMD with symptoms of orofacial pain and limited range of jaw opening.

Exclusion Criteria:

* Previous head, neck or TMJ traumas.
* History of temporomandibular joint surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Anamnestic questionnaire by Fonseca | Baseline (pre-treatment), 3rd and week 7 (post-treatment)
  To evaluate TMD by 10 questions with their corresponding scores from 0 to 10
Craniocervical angle - CVA | Baseline (pre-treatment), 3rd and week 7 (post-treatment)
  photographic method to evaluate the angle where an angle less than 50 degrees will be considered as forward head posture

SECONDARY OUTCOMES:
Boley Gauge | Baseline (pre-treatment), 3rd and week 7 (post-treatment)
  Electronic Digital Caliper to assess mouth opening (active/passive)
Visual Analog Scale (VAS) | Baseline (pre-treatment), 3rd and week 7 (post-treatment)
  0-10 scale (zero represents no pain and 10 is the worst pain ever) to record orofacial pain
Mandibular Opening | Baseline (pre-treatment), 3rd and week 7 (post-treatment)
  Tape to measure the distance between the incisal edges of upper and lower teeth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Lee WY, Okeson JP, Lindroth J. The relationship between forward head posture and temporomandibular disorders. J Orofac Pain. 1995 Spring;9(2):161-7. PMID 7488986
- [Background] Salkar RG, Radke UM, Deshmukh SP, Radke PM. Relationship between temporomandibular joint disorders and body posture. Int J Dent Health Sci. 2015;2(6):1523-30.
- [Background] Saddu SC, Dyasanoor S, Valappila NJ, Ravi BV. The Evaluation of Head and Craniocervical Posture among Patients with and without Temporomandibular Joint Disorders- A Comparative Study. J Clin Diagn Res. 2015 Aug;9(8):ZC55-8. doi: 10.7860/JCDR/2015/12830.6343. Epub 2015 Aug 1. PMID 26436048
- [Background] El-Hamalawy FA. Forward head correction exercises for management of myogenic tempromandibular joint dysfunction. 2011;7(8)
- [Background] Tang Y, Xu LL, Fan S. [Control study of forward head posture between patients with temporomandibular disorders and healthy people]. Shanghai Kou Qiang Yi Xue. 2021 Apr;30(2):173-176. Chinese. PMID 34109357
- [Background] Xiao CQ, Wan YD, Li YQ, Yan ZB, Cheng QY, Fan PD, Huang Y, Wang XY, Xiong X. Do Temporomandibular Disorder Patients with Joint Pain Exhibit Forward Head Posture? A Cephalometric Study. Pain Res Manag. 2023 Feb 2;2023:7363412. doi: 10.1155/2023/7363412. eCollection 2023. PMID 36776487
- [Background] Minervini G, Franco R, Marrapodi MM, Crimi S, Badnjevic A, Cervino G, Bianchi A, Cicciu M. Correlation between Temporomandibular Disorders (TMD) and Posture Evaluated trough the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD): A Systematic Review with Meta-Analysis. J Clin Med. 2023 Apr 2;12(7):2652. doi: 10.3390/jcm12072652. PMID 37048735